CLINICAL TRIAL: NCT04850547
Title: Vitamin D Status and Bone Turnover Markers in Patients With Non Alcoholic Fatty Liver Disease
Brief Title: Effect of Fatty Liver Disease on Bone Density
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samar Hussein Kamel, Assistant lecturer at tropical medicine and gastroenterology, Sohag University
Other Study IDs: IRB00013006
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Osteoporosis
Keywords: Non Alcoholic Fatty Liver osteocalcin osteoporosis vitamin D
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Non Alcohlic Fatty Liver (NAFLD) is a spectrum of diseases that ranges from accumulation of fat in the liver (Hepatosteatosis) that may be accompanied by inflammation (Steatohepatitis) to necrosis, fibrosis and even cirrhosis resembling alcoholic hepatitis in the absence of alcoholic abuse (Pardee et al., 2012).

It has been estimated that the global prevalence of NAFLD is as high as one billion. In the United States, NAFLD is estimated to be the most common cause of chronic liver disease, affecting between 80 and 100 million individuals, among whom nearly 25% progress to NASH (Loomba et al., 2013).

In general, the prevalence of NAFLD has increased over the last 20 years. The Middle East and South America have the highest NAFLD prevalence at 31% and 32% respectively with the lowest prevalence in Africa at 13.5% (Younossi et al., 2016).

Liver biopsy (LB) is still the standard test of NAFLD diagnosis and the presence of early liver fibrosis. However, histologic lesions are not evenly distributed throughout the liver. A sampling error is the biggest limitation in the diagnosis of NAFLD by LB with inflammatory lesions and ballooning degeneration potentially resulting in misdiagnoses and staging inaccuracies (Lee et al., 2016).

To overcome these limitations, several non-invasive markers have been used instead of liver biopsy. These methods are either laboratory markers or imaging modalities. Controlled attenuation parameter (CAP) is a new technology based on the principle of the ultrasonic attenuation of transient elastography depending on the viscosity [fat] of the medium [liver] and the distance of propagation of the ultrasonic signals into the liver, providing a useful method for the quantitative detection of liver fat content and is considered a better assessment method for hepatic steatosis. Compared with ultrasound, this technology improves the sensitivity and specificity for the diagnosis of fatty liver and can be used for universal screening, diagnosis, and follow-up in NAFLD patients (Sasso et al., 2016).

NAFLD is known to be closely associated with metabolic conditions, including insulin resistance, abdominal obesity, dyslipidaemia and type 2 diabetes, and is thus regarded as the hepatic manifestation of the metabolic syndrome (Ballestri., 2016). In recent epidemiological studies, NAFLD was shown to be connected with diseases that are usually not dependent on obesity, such as sarcopenia and osteoporosis (Poggiogalle et al., 2017).

Osteoporosis is becoming a public health problem all over the world. Disability resulting from low-energy fractures, e.g: hip or vertebral fractures, is the major concern for early detection and treatment. It is estimated that osteoporosis affects 200 million women worldwide (Kanis et al., 2007).

Liver is the source of many proteins and is the regulator of several pathways involving bone metabolism; one of the most well-known of all is vitamin D metabolism pathway. Considering the role of liver in bone metabolism, the association between NAFLD and bone abnormalities is not surprising especially with substantial supporting evidences in recent years (Eshraghian et al., 2017).

Besides its role in the calcium and bone metabolism, vitamin D may also exert pleiotropic effects in many tissues. NAFLD patients were reported to have a marked reduction in serum 25(OH) vitamin D when compared with controls (Yilmaz et al., 2011).

In adults, bone is constantly being remodeled, first being broken down (bone resorption) and then being rebuilt (bone formation). The resorption and reformation of bone is important for repair of microfractures and to allow modification of structure in response to stress and other biomechanical forces. Bone formation is normally tightly coupled to bone resorption, so that bone mass does not change. Bone diseases occur when formation and resorption are uncoupled. Several assays are available that measure bone turnover markers (BTMs). These assays measure collagen breakdown products and other molecules released from osteoclasts and osteoblasts during the process of bone resorption and formation. Markers that are specific to bone formation include bone-specific alkaline phosphatase (BSAP), osteocalcin, and N-terminal propeptide of type I procollagen (PINP); markers specific to bone resorption include N-terminal telopeptide of type I collagen (NTX), C-terminal telopeptide of type I collagen (CTX), and pyridinoline cross-links (Rosen et al., 2019).

DETAILED DESCRIPTION:
All included patients will be subjected to the following:

1. Complete history taking including age, sex, current medical history (e.g. hypertension, diabetes mellitus, cardiovascular disease, renal, thyroid, parathyroid diseases and menopausal status), daily alcohol consumption and smoking status will be recorded from interviews with the participants during the examination.
2. thorough clinical examination. The participants' anthropometric measurements will be obtained including: their body weight, height, waist circumference (WC) and body mass index (BMI).

   General examination Arterial blood pressure will be recorded and for detection of stigmata of chronic liver disease.

   Abdominal examination will be done for assessment of the size of the liver and spleen.
3. Diagnosis of NAFLD:

   The diagnosis will be based on abdominal ultrasound findings and will be confirmed by fibroscan examination as the following:
   1. Abdominal ultrasound: steatosis will be graded according to Quinn and Gosink (1985) as the following:

      Grade I: Minimal diffuse increase in the fine echoes. Liver appears bright compared to the cortex of the kidney.

      Grade II: Moderate diffuse increase in the fine echoes. Slightly impaired visualization of the intrahepatic vessels and diaphragm.

      Grade III: Marked increase in the fine echoes. Poor or no visualization of intrahepatic vessels and diaphragm and poor penetration of the posterior segment of the right lobe of the liver
   2. Fibosscan to evaluate steatosis grades by CAP score and fibrosis stages as described by (Sasso et al., 2010).
4. Laboratory investigations:

   1. Complete Blood Count (CBC).
   2. Liver profile: alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum albumin, total and direct bilirubin, prothrombin time and INR.
   3. Renal profile: creatinine and urine analysis.
   4. Total cholesterol, triglyceride (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C).
   5. Fasting blood sugar.
   6. (HBsAg, HCV Ab) Viral markers.
   7. 25-hydroxyl-vitamin D (25(OH)D) in serum.
   8. Serum Osteocalcin as a marker of bone formation and serum NTX as a marker of bone resorption.

ELIGIBILITY:
Inclusion Criteria:

* Males (20-60 years old ) and premenopausal females with NAFLD diagnosed by Fibroscan

Exclusion Criteria:

* (i) Patients aged <20 years or >60years. (ii) Alcohol consumption of ≥30 g/day in men or≥20 g/day in women. (iii) Subjects with suspected or proven any other liver disease other than NAFLD as (viral hepatitis, drug-induced liver injury, autoimmune liver disease, Wilson's disease or primary biliary cholangitis).

(iv) Postmenopausal females to avoid the increased risk of osteoporosis in those patients due to hormonal changes.

(v) Patients with conditions known to affect bone metabolism, such as kidney, thyroid or parathyroid diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects (attending either the Tropical Medicine and Gastroenterology Outpatient Clinic or the Inpatient section of the department) will be recruited from male and premenopausal female patients suffering from dyspeptic symptoms and underwent routine abdominal ultrasound which revealed bright liver.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
level of serum 25(OH) vitamin D in NAFLD patients patients | A year
  • To study level of serum 25(OH) vitamin D in NAFLD patients and its relationship to disease severity.
level of osteocalcin in NAFLD patients | A year
  • To study serum level of osteocalcin and (marker of bone formation) and NTX(marker of bone resorption) in NAFLD patients.
Correlation between bone and liver | A year
  To assess the correlation between bone turnover markers and liver steatosis and fibrosis in NAFLD patients

CONTACTS AND LOCATIONS:
Overall Officials: Samar Hussein, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poggiogalle E, Donini LM, Lenzi A, Chiesa C, Pacifico L. Non-alcoholic fatty liver disease connections with fat-free tissues: A focus on bone and skeletal muscle. World J Gastroenterol. 2017 Mar 14;23(10):1747-1757. doi: 10.3748/wjg.v23.i10.1747. PMID 28348479
- [Background] Ballestri S, Zona S, Targher G, Romagnoli D, Baldelli E, Nascimbeni F, Roverato A, Guaraldi G, Lonardo A. Nonalcoholic fatty liver disease is associated with an almost twofold increased risk of incident type 2 diabetes and metabolic syndrome. Evidence from a systematic review and meta-analysis. J Gastroenterol Hepatol. 2016 May;31(5):936-44. doi: 10.1111/jgh.13264. PMID 26667191
- [Background] Eshraghian A. Bone metabolism in non-alcoholic fatty liver disease: vitamin D status and bone mineral density. Minerva Endocrinol. 2017 Jun;42(2):164-172. doi: 10.23736/S0391-1977.16.02587-6. Epub 2016 Dec 14. PMID 27973461
- [Background] Sasso M, Audiere S, Kemgang A, Gaouar F, Corpechot C, Chazouilleres O, Fournier C, Golsztejn O, Prince S, Menu Y, Sandrin L, Miette V. Liver Steatosis Assessed by Controlled Attenuation Parameter (CAP) Measured with the XL Probe of the FibroScan: A Pilot Study Assessing Diagnostic Accuracy. Ultrasound Med Biol. 2016 Jan;42(1):92-103. doi: 10.1016/j.ultrasmedbio.2015.08.008. Epub 2015 Sep 19. PMID 26386476
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- See also: Related Info — http://www.uptodate.com.